CLINICAL TRIAL: NCT07047729
Title: COMPARATIVE OUTCOME OF EARLY AND STANDARD ORAL FEEDING AFTER EMERGENCY BOWEL SURGERY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Hamail Khanum (Other)
Responsible Party: Sponsor-Investigator, Dr Hamail Khanum, Consultant, Gulab Devi Hospital
Organization: Gulab Devi Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Bowel Surgery; Emergency Abdominal Surgery; ERAS

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A with early oral feeding (ERAS) (Experimental): Group A (early oral feeding), consisting of 30 patients. In Group A, a liquid diet will be initiated within 24 hours after surgery and, if well-tolerated without vomiting, will transition to a regular diet over the subsequent 24 hours. Tolerance to oral feeding will be evaluated by monitoring for vomiting within the first 24 hours after initiating a regular diet. Patients will be discharged from the hospital once they have tolerated a regular diet for at least 24 hours and the duration of hospital stay will be noted as well.
  Interventions: Other: Early oral feeding
- Group B with standard oral feeding (Experimental): Group B (standard oral feeding), consisting of 30 patients. A standard diet (late feeding), including liquid filtrates, will only be introduced after the resolution of the ileus, during which these patients will remain NPO (nothing by mouth). Tolerance to oral feeding will be evaluated by monitoring for vomiting within the first 24 hours after initiating a regular diet. Patients will be discharged from the hospital once they have tolerated a regular diet for at least 24 hours and the duration of hospital stay will be noted as well.
  Interventions: Other: Standard oral feeding

INTERVENTIONS:
Other: Early oral feeding — Liquid diet will be initiated within 24 hours after surgery and, if well-tolerated without vomiting, will transition to a regular diet over the subsequent 24 hours
  Arms: Group A with early oral feeding (ERAS)
Other: Standard oral feeding — Standard diet (late feeding), including liquid filtrates, will only be introduced after the resolution of the ileus, during which these patients will remain NPO (nothing by mouth).
  Arms: Group B with standard oral feeding

SUMMARY:
Informed consent will be obtained from patients or their legal representatives in cases where the patient is unconscious. Patient information, including names, ages, gender, smoking history, comorbidities, and the indication for emergency surgical procedures, will be documented. All surgical procedures will follow standard protocols and will be conducted by a single surgical team led by at least two consultants, each with more than five years of experience. All 60 patients will be randomly allocated into two groups using a random number table: Group A (early oral feeding), consisting of 30 patients, and Group B (standard oral feeding), consisting of 30 patients. In Group A, a liquid diet will be initiated within 24 hours after surgery and, if well-tolerated without vomiting, will transition to a regular diet over the subsequent 24 hours. On the other hand, in Group B, a standard diet (late feeding), including liquid filtrates, will only be introduced after the resolution of the ileus, during which these patients will remain NPO (nothing by mouth).

DETAILED DESCRIPTION:
Informed consent will be obtained from patients or their legal representatives in cases where the patient is unconscious. Patient information, including names, ages, gender, smoking history, comorbidities, and the indication for emergency surgical procedures, will be documented. All surgical procedures will follow standard protocols and will be conducted by a single surgical team led by at least two consultants, each with more than five years of experience. All 60 patients will be randomly allocated into two groups using a random number table: Group A (early oral feeding), consisting of 30 patients, and Group B (standard oral feeding), consisting of 30 patients. In Group A, a liquid diet will be initiated within 24 hours after surgery and, if well-tolerated without vomiting, will transition to a regular diet over the subsequent 24 hours. On the other hand, in Group B, a standard diet (late feeding), including liquid filtrates, will only be introduced after the resolution of the ileus, during which these patients will remain NPO (nothing by mouth). Tolerance to oral feeding will be evaluated by monitoring for vomiting within the first 24 hours after initiating a regular diet, and this evaluation will be conducted by the researcher herself. Patients will be discharged from the hospital once they have tolerated a regular diet for at least 24 hours and the duration of hospital stay will be noted as well. All data will be documented on a predefined proforma. Other variables like febrile episode and need for additional NPO will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Either Gender
* Requiring emergency surgery due to conditions such as obstructive bowel disease, GI perforation, colorectal surgery, blunt abdominal trauma (resulting from falls or roadside accidents), and penetrating abdominal trauma (involving firearm injuries and stab wounds).

Exclusion Criteria:

* Patients with terminal cancer need palliative surgery (as their focus is on comfort care rather than surgical intervention).
* Patients who had undergone surgery within the past 30 days (to avoid potential complications associated with recent surgical procedures).
* Patients receive regular renal replacement therapy (to prevent additional stress on their medical condition).
* Pregnant women (as surgical interventions may pose risks to both the mother and the unborn child).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2025-09-06 (Estimated); Study Completion 2025-09-06 (Estimated)

PRIMARY OUTCOMES:
Hospital stay | 10 Days
  Duration from day of surgery till discharge following discharge criteria
Feed tolerance | 24 hours
  Tolerance to oral feeding will be evaluated by monitoring for vomiting within the first 24 hours after initiating a regular diet

CONTACTS AND LOCATIONS:
Overall Officials: Professor Dr Maratab Ali, MBBS FCPS, Study Director — Gulab Devi Hospital
Locations (1):
- Gulab Devi Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No